CLINICAL TRIAL: NCT06531005
Title: Assessment of Ventilation Parameters for Extubation Prediction in ICU
Status: Recruiting | Type: Observational
Sponsor: Ankara University (Other)
Collaborators: Gazi University (Other)
Responsible Party: Principal Investigator, Nuri Isler, Research assistant, Ankara University
Other Study IDs: Respmechanics
Record Dates: First submitted 2024-07-24; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Acute Respiratory Failure; Invasive Mechanical Ventilation
Keywords: respiratory failure; extubation; mechanical power; elastic power; repiratory mechanics; outcome
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to research the values of mechanical power, driving pressure, and elastic power in predicting the duration of mechanical ventilation in critically ill patients undergoing invasive mechanical ventilation. This will help determine which patients may be considered for early extubation, which patients should wait for extubation, and the patients where extubation is anticipated to be prolonged, attention should be paid to initiating preparations for alternative treatment methods like tracheostomy early.

DETAILED DESCRIPTION:
Due to acute respiratory failure, mechanical ventilation support is provided to over 20 million patients worldwide. Therefore, various studies are being conducted to prevent ventilation-associated lung injury in patients receiving invasive mechanical ventilation, especially in conditions such as acute respiratory distress syndrome (ARDS).

Initially, protective mechanical ventilation studies have shown that keeping plateau pressure (Pplat), reflecting static compliance, below 30 cmH2O along with low tidal volume reduces all-cause mortality. Subsequent studies have defined driving pressure as Pplato-PEEP, suggesting that keeping driving pressure below 15 cmH2O may reduce excessive strain on healthy lung tissue and the development of ventilator-associated lung injury.

In 2016, Gattinoni and colleagues defined mechanical power as the power applied by the ventilator to the entire respiratory system per minute during mechanical ventilation, prompting research into the relationship between mechanical power and mortality, particularly in ARDS.

Mechanical power consists of three components: energy delivered with each breath when PEEP is applied, energy applied to overcome airway resistance, and elastic energy delivered with each tidal breath.

Finally, Yongpeng Xie and colleagues hypothesized that elastic power, normalized by compliance, has a more significant relationship with mortality in ARDS patients. Studies on mechanical power, driving pressure, and elastic power typically focus on values measured on the first day of intubation and are predominantly conducted in ARDS patients.

By including all patients under invasive mechanical ventilation in the study, the importance of measuring and monitoring mechanical ventilator parameters (mechanical power, driving pressure, and elastic power) at 0th, 24th, and 48th hours to predict extubation within the first week is being determined. This aims to identify when early extubation should be considered, when extubation should be delayed, and to prepare for alternative treatment options like tracheostomy in cases where extubation might be prolonged.

ELIGIBILITY:
Inclusion Criteria:

* consenting patients who have recently been intubated for acute respiratory failure

Exclusion Criteria:

* patients with lung cancer/ lung metastasis
* ECMO
* death within 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who have recently been intubated for acute respiratory failure and admitted to participating ICUs will be screened and included in the study if eligible.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
extubation time | seven days
  time patients will be extubated after intubation

SECONDARY OUTCOMES:
mortality | 28 days
  28 day mortality
acute renal failure | one month
  Number of patients who developed acute kidney injury according to KDIGO guidelines
ICU/ hospital length of stay | three months
  ICU/ hospital length of stay

CONTACTS AND LOCATIONS:
Overall Officials: Neriman D Altıntaş, Professor, Principal Investigator — https://avesis.ankara.edu.tr/ndaltintas
Locations (1):
- Ankara University Faculty of Medicine, Altindağ, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Adhikari NK, Fowler RA, Bhagwanjee S, Rubenfeld GD. Critical care and the global burden of critical illness in adults. Lancet. 2010 Oct 16;376(9749):1339-46. doi: 10.1016/S0140-6736(10)60446-1. Epub 2010 Oct 11. PMID 20934212
- [Background] Acute Respiratory Distress Syndrome Network; Brower RG, Matthay MA, Morris A, Schoenfeld D, Thompson BT, Wheeler A. Ventilation with lower tidal volumes as compared with traditional tidal volumes for acute lung injury and the acute respiratory distress syndrome. N Engl J Med. 2000 May 4;342(18):1301-8. doi: 10.1056/NEJM200005043421801. PMID 10793162
- [Background] de Durante G, del Turco M, Rustichini L, Cosimini P, Giunta F, Hudson LD, Slutsky AS, Ranieri VM. ARDSNet lower tidal volume ventilatory strategy may generate intrinsic positive end-expiratory pressure in patients with acute respiratory distress syndrome. Am J Respir Crit Care Med. 2002 May 1;165(9):1271-4. doi: 10.1164/rccm.2105050. PMID 11991877
- [Background] Amato MB, Meade MO, Slutsky AS, Brochard L, Costa EL, Schoenfeld DA, Stewart TE, Briel M, Talmor D, Mercat A, Richard JC, Carvalho CR, Brower RG. Driving pressure and survival in the acute respiratory distress syndrome. N Engl J Med. 2015 Feb 19;372(8):747-55. doi: 10.1056/NEJMsa1410639. PMID 25693014
- [Background] Marini JJ, Rocco PRM, Gattinoni L. Static and Dynamic Contributors to Ventilator-induced Lung Injury in Clinical Practice. Pressure, Energy, and Power. Am J Respir Crit Care Med. 2020 Apr 1;201(7):767-774. doi: 10.1164/rccm.201908-1545CI. PMID 31665612
- [Result] Gattinoni L, Tonetti T, Cressoni M, Cadringher P, Herrmann P, Moerer O, Protti A, Gotti M, Chiurazzi C, Carlesso E, Chiumello D, Quintel M. Ventilator-related causes of lung injury: the mechanical power. Intensive Care Med. 2016 Oct;42(10):1567-1575. doi: 10.1007/s00134-016-4505-2. Epub 2016 Sep 12. PMID 27620287
- [Result] Xie Y, Yan Y, Shi J, Luo J, Wang Y, Chen H, Li X. Elastic power, a novel predictor of the severity and prognosis of ARDS. J Crit Care. 2023 Dec;78:154380. doi: 10.1016/j.jcrc.2023.154380. Epub 2023 Jul 20. PMID 37480658